CLINICAL TRIAL: NCT00480402
Title: Eficacia de Los Suplementos de Progesterona Natural en la prevención Del Parto pretérmino Gemelar
Brief Title: Natural Progesterone and Preterm Birth in Twins
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VLC-VS-0405-507-23
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Preterm Birth
Keywords: preterm birth; progesterone; twins; Preterm birth in twin gestations
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 400 mg Progesterone (Experimental): Approximately one third of the bichorionic biamniotic twin pregnant women randomized to the 400 mg Progesterone Group vaginal pessaries arm.
  Interventions: Drug: 400 mg Progesterone
- 200 mg Progesterone Group (Experimental): Approximately one third of the bichorionic biamniotic twin pregnant women randomized to the 200 mg Progesterone Group vaginal pessaries arm.
  Interventions: Drug: 200 mg of Progesterone
- Placebo (Active Comparator): Approximately one third of the bichoronic biamniotic twin pregnant women were randomized to the placebo vaginal pessaries arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 200 mg of Progesterone — Administration of 200 mg of Progesterone
  Arms: 200 mg Progesterone Group
Drug: 400 mg Progesterone — Administration of 400 mg Progesterone
  Arms: 400 mg Progesterone
Drug: Placebo — Administration of a Placebo
  Arms: Placebo

SUMMARY:
To assess the effectiveness of natural progesterone supplementation in preventing preterm births in twins.

DETAILED DESCRIPTION:
Objective: To assess the effectiveness of natural progesterone supplementation in preventing preterm births in twins.

Study Design: National multicenter randomized double blind controlled clinical trial.

Setting: Six tertiary hospitals in the east of Spain (communities of Valencia and Murcia): Instituto Universitario IVI Valencia, Hospital Universitario La Fe (Valencia), Hospital Universitario Dr. Peset (Valencia), Hospital General Universitario (Alicante), Hospital Vega Baja de Orihuela (Alicante) y Hospital Virgen de la Arrixaca (Murcia).

Population: 246 bichorionic biamniotic twin pregnant women divided in three groups according to the allocated randomized treatment: (I) placebo (N=82); (II) 200 mg progesterone (N=82); and (III) 400 mg progesterone (N=82).

Methods: All participant women will self-administer two vaginal pessaries at bedtime containing the allocated treatment. Vaginal pessaries will be identical externally but will contain either placebo or 200 mg of natural progesterone (Laboratorios Effik, Madrid, Spain). The treatment will be applied from the 20th week until the 34th week (or until delivery if it occurred earlier). Control visits will be performed at 24, 28, 32 and 34 weeks. Pregnancies will be managed according to each local protocol. An external statistical analysis will be performed on intention to treat basis.

Main outcome measure: Preterm birth rate (<37 weeks). Secondary outcome measures: very preterm birth rate (<32 weeks); cervical length measured by vaginal ultrasound at each control visit; need for tocolytic treatments; rate of preterm premature rupture of membranes; and perinatal morbidity and mortality.

Estimated period of study: 2006-2008.

ELIGIBILITY:
Inclusion Criteria:

* Bichorionic biamniotic twin pregnant women
* = or > 18 years old

Exclusion Criteria:

* Single pregnancy or monochorionic twin pregnancy or triplets
* Chronic hepatic pathology, previous alterations in hepatic analysis during anti-contraceptive treatment; or gestational cholestasis in in previous pregnancies.Basal alterations in hepatic analysis profile.
* Profylactic cerclage until week 14.
* Basal alterations in renal analysis profile
* Local allergy to micronized natural progesterone
* Genital pathology not allowing for correct absorption of medication
* Fetal anomoly diagnosed after sonograph week 12 and/or 20.
* Smokers of more than 10 cigarettes/day
* Consumers of illegal substances

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Serra, MDPhD, Study Director — Instituto Valenciano de la Infertilidad
Locations (1):
- Instituto Valenciano de la Infertilidad, Valencia, Valencia, Spain